CLINICAL TRIAL: NCT02888132
Title: Echocardiography-guided Transthoracic Radio Frequency/Laser Ablation for Ventricular Septum of Hypertrophic Obstructive Cardiomyopathy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KY20162042-1
Record Dates: First submitted 2016-08-29; First posted 2016-09-02 (Estimated); Last update posted 2016-09-02 (Estimated); Status verified 2016-08

CONDITIONS: Hypertrophic Obstructive Cardiomyopathy
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic

ARMS (1):
- Hypertrophic Obstructive Cardiomyopathy (Experimental)
  Interventions: Procedure: Echocardiography-guided transthoracic radio frequency ablation for HOCM ventricular septum; Procedure: Echocardiography-guided transthoracic laser ablation for HOCM ventricular septum

INTERVENTIONS:
Procedure: Echocardiography-guided transthoracic radio frequency ablation for HOCM ventricular septum
Procedure: Echocardiography-guided transthoracic laser ablation for HOCM ventricular septum

SUMMARY:
Hypertrophic Obstructive Cardiomyopathy (HOCM) patients have significant clinical symptoms, including progressively increasing fatigue, angina, exertional dyspnea, and syncope. Conservative medications are used to treat the vast majority of patients. Invasive therapy, which includes surgical myectomy, septal ethanol ablation and dual-chamber pacing is introduced to patients with refractory symptoms or drug resistance. Considering the sternotomy and relatively high patients' tolerance required in myectomy, the potentially risky misplacement of ethanol and the anatomic variability of the vascularised hypertrophic septum, and the potential risk of conduction block after these two treatments, the development of new minimally invasive approach is warranted.

Previous researches have illustrated the effectiveness and feasibility of transcatheter radio frequency ablation for HOCM patients. By far, there has been no report on transthoracic laser-induced interstitial thermotherapy (LITT) for human treatment. Since 2004, our department has adopted High Intensity Focused Ultrasound, radio frequency and laser in solid tumors treatment, including liver tumors and fibroid. Also our center has conducted several animal experiments to verify the feasibility of radio frequency/laser in septal myocardium ablation.

The purpose of this study is to lead echocardiography-guided transthoracic radio frequency/laser ablation for HOCM ventricular septum, make minimally invasive treatment plans for HOCM patients, and verify the safety and validity of intervention treatment in long term.

ELIGIBILITY:
Inclusion Criteria:

* Subject who cannot tolerate ventricular septum resection or transcatheter ethanol ablation and volunteer for the operation
* Subject meets HOCM diagnosis standards verified by the echocardiogram; the obstruction is located in the basal part of ventricular septum
* Subject has significant clinical symptoms, including progressively increasing fatigue, angina, exertional dyspnea, and syncope; subject receives poor effect after drug therapy or cannot tolerate side effects of medication
* Subject has pressure gradient of left ventricular outflow tract (LVOT) ≥50 mmHg（with Systolic Anterior Motion）in the resting-state or after exercise stress test
* Subject over 18 years old

Exclusion Criteria:

* Subject has non-obstructive hypertrophic cardiomyopathy
* Subject has combined cerebral vascular diseases
* Subject has diseases that must receive surgeries, including severe mitral valve lesions and coronary heart disease which requires coronary artery bypass grafting.
* Subject has end-stage heart failure
* Subject has intraventricular septal thickness (IVST) ≥ 30mm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2016-04; Primary Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
Mortality | 24 months
Quantification of obstructive severity | 24 months
  Investigators use pressure gradient of left ventricular outflow tract (LVOT) to quantify obstructive severity. If the pressure gradient increases, the symptom gets deteriorated; if the pressure gradient decreases, the symptom gets relieved.

SECONDARY OUTCOMES:
Quantification of cardiac function | 24 months
  Investigators use ejection function (EF) to quantify the systolic function. If EF is higher after the operation, the systolic function gets improved; if EF lower after the operation, the systolic function gets deteriorate. Investigators use diastolic degree to evaluate the diastolic function. If diastolic degree is lower after the operation, the diastolic function gets improved; If diastolic degree is higher after the operation, the diastolic function gets deteriorated.
Quantification of conduction block | 24 months
  If there is no conduction block observed, the therapy is successful; if there is conduction block, it could be considered as one potential complication.

CONTACTS AND LOCATIONS:
Locations (1):
- Ultrasound Medicine Department of Xijing Hospital, Fourth Military Medical University, Xi'an, Shaanxi, China

REFERENCES:
- [Derived] Ta S, Li J, Hsi DH, Hu R, Lei C, Shan B, Li W, Wang J, Wang B, Kang N, Li X, Liu J, Qi C, Huang J, Han Y, Ruan F, Zhang J, Liu L. Percutaneous intramyocardial septal radiofrequency ablation after 5-year follow-up. Heart. 2024 May 10;110(11):792-799. doi: 10.1136/heartjnl-2023-323606. PMID 38388470
- [Derived] Wang XY, Wang B, Zhu XL, Ma ZL, Liu Y, Lei CH, Yang QL, Hu D, Zhao XL, Liu ZR, Liu LW. Clinical and molecular characterization of seven patients with Danon disease. Exp Ther Med. 2021 Apr;21(4):395. doi: 10.3892/etm.2021.9826. Epub 2021 Feb 24. PMID 33680117